CLINICAL TRIAL: NCT05840237
Title: REGAIN: A Randomized, Double Blind, Placebo Controlled Trial to Determine the Effects of Oxaloacetate on Improving Fatigue in Long COVID
Brief Title: REGAIN: RCT of Oxaloacetate for Fatigue in Long COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terra Biological LLC (Industry)
Collaborators: Bateman Horne Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TB-2023-AEO LC
Record Dates: First submitted 2023-04-28; First posted 2023-05-03 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-11

CONDITIONS: Post-COVID-19 Syndrome; Fatigue Syndrome, Chronic
Keywords: Long COVID; COVID; Fatigue; Oxaloacetate; COVID Fatigue
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Fatigue Syndrome, Chronic; Fatigue | interventions — Oxaloacetic Acid; Flour

STUDY DESIGN:
Intervention Model Description: Single Center, Randomized, Placebo Controlled, Double Blind
Who Masked: Participant, Care Provider, Investigator
Masking Description: Individual patients will be randomized, and will receive a numbered bottle that corresponds to either Oxaloacetate or placebo. At the end of the trial, the blind will be broken to reveal which participant is in which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxaloacetate Arm (Experimental): 1,000 mg of Anhydrous Enol-Oxaloacetate taken BID with Breakfast and Lunch
  Interventions: Other: Anhydrous Enol-Oxaloacetate, a "Medical Food"
- Placebo Arm (Placebo Comparator): 1,000 mg of white Rice Flour taken BID with Breakfast and Lunch
  Interventions: Other: White Rice Flour

INTERVENTIONS:
Other: Anhydrous Enol-Oxaloacetate, a "Medical Food" — Treatment with the medical food "Oxaloacetate CFS", 2 - 500 mg capsules BID with food
  Other Names: Oxaloacetate, Oxaloacetate CFS
  Arms: Oxaloacetate Arm
Other: White Rice Flour — Treatment with the food "White Rice Flour", 2- 500 mg capsules BID with food
  Other Names: Rice Flour
  Arms: Placebo Arm

SUMMARY:
Following acute COVID-19, some patients develop a group of debilitating symptoms that include fatigue, orthostatic intolerance, difficulty with attention and concentration (often called "brain fog"), myalgias and disrupted sleep. The term Long COVID is used to describe these symptoms after the initial viral infection has passed. These symptoms are the same as those that define myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS).

A "Proof of Concept" trial showed significant fatigue benefit in Long COVID patients. This randomized, placebo controlled follow-on trial will determine whether oxaloacetate can reduce fatigue and improve other symptoms in patients with Long COVID who meet diagnostic criteria for ME/CFS.

DETAILED DESCRIPTION:
Following acute COVID-19, some patients develop a group of debilitating symptoms that include fatigue, orthostatic intolerance, difficulty with attention and concentration (often called "brain fog"), myalgias and disrupted sleep (1-8). The term Long COVID is used to describe the prolonged multisystem illness that occurs after acute infection with SARS-CoV-2. The frequency with which this syndrome occurs following acute COVID-19 ranges from 2-40% of cases (8, 9). Although individuals with more severe acute COVID-19 are more likely to develop Long COVID, it is prevalent in people who were mildly symptomatic or asymptomatic at the time of acute infection with SARS-CoV-2 (8, 10, 11).

Many people with Long COVID remain ill for many months. Currently there are thousands of people in the U.S. that have been suffering with Long COVID for the past three years since the onset of the COVID-19 pandemic in January 2020 (12). In a recent study, the Imperial College in London estimated that there are 2 million adults suffering from Long COVID in the UK (13). According to the US News, Long COVID has become the 'Pandemic After the Pandemic (14). There is evidence that diagnosis and treatment early in the course of illness improves the likelihood of recovery and sustained remission of post-infectious illness (15, 16).

A code U09.9 was added to ICD-10 in October 2021 to document post-acute sequela of COVID-19 after infection and Long COVID. The WHO published a Long COVID clinical case definition coincident with the ICD code that described the common symptoms of Long COVID including fatigue, shortness of breath, cognitive dysfunction but also others and these generally have an impact on everyday functioning (17). The signs and symptoms described in this case definition were also described in survey responses from an international cohort of more than 6,000 people with Long COVID (18). This study found that signs and symptoms that persisted more than 6 months of illness included fatigue, brain fog, post-exertional malaise, insomnia, joint and muscle pain, orthostatic intolerance, gastrointestinal symptoms, and sensorimotor symptoms including tremors and nerve pain. These symptoms are the same as those that define myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). ME/CFS is defined by the National Academy of Medicine as a substantial reduction or impairment in the ability to engage in pre-illness levels of activity (occupational, educational, social, or personal life) that lasts for more than 6 months and is accompanied by profound fatigue of new onset that is not a result of ongoing or unusual excessive exertion and is not alleviated by rest; post-exertional malaise (PEM) which is the worsening of symptoms after physical, mental, or emotional exertion that would not have caused a problem before the illness; unrefreshing sleep; and at least one of the following two additional manifestations must be present, cognitive impairment or orthostatic intolerance (18).

Oxaloacetate is an energy metabolite found in every cell of the human body. It holds a key place in the TCA cycle within the mitochondria, providing energy to the cells. It is also a critical early metabolite in gluconeogenesis, which provides glucose for the heart and brain during times of low glucose. In addition, oxaloacetate is found in the urea cycle (which converts toxic ammonia to urea), amino acid synthesis, and fatty acid synthesis. It is critical to human metabolism and proper cellular function, and it is central to energy production and use in the body.

A "Proof of Concept" trial showed significant fatigue benefit in Long COVID patients. This randomized, placebo controlled follow-on trial will determine whether oxaloacetate can reduce fatigue and improve other symptoms in patients with Long COVID who meet diagnostic criteria for ME/CFS.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form. Male or female, 18 to 65 years of age. Able to read, understand and voluntarily sign the informed consent form.

Diagnosed with Long COVID by a provider after suspected, probable or confirmed infection with SARS-CoV-2 as defined by the WHO (see full protocol for details). Patients have experienced moderate to severe fatigue at least 50% of the time over the past 6 months that is not relieved by rest and post-exertional malaise (PEM) which is unusual worsening of symptoms after minimal physical or cognitive exertion, which can occur or persist 24 hours or more after the exertion.

Agree to refrain from taking medications that would affect assessment of the effectiveness of study IP for the duration of the study.

Females of childbearing potential should be on adequate contraception such as oral, implantable, injectable or transdermal hormonal contraceptives (should have been used for a minimum of one full cycle prior to administration of study drug), intrauterine devices (IUD), vasectomized partner, double barrier method (male or female condom, sponge, diaphragm or vaginal ring with simultaneous use of spermicidal jelly or cream).

Each patient of child-bearing potential must have a negative urine pregnancy test at Visit 1. The urine test at Visit 1 must be confirmed negative prior to dispensing IP. Women of child-bearing potential will have a urine pregnancy test at each visit (2 and 3) and it must be negative to continue. Women who are confirmed to be of non-childbearing potential do not require pregnancy testing. To be considered of non-child-bearing potential, the patient must be: post-menopausal (defined as no menses for at least one year); or surgically sterile (s/p hysterectomy, bilateral oophorectomy or bilateral tubal ligation at least 6 months prior to randomization); or at least 3 months s/p a non-surgical permanent sterilization procedure.

Stated willingness to comply with all study procedures. Be available and appear for the 3 in-person visits of the study. Have mobile (smart) phone and access to the internet. Willingness to wear a device on their ankle.

Exclusion Criteria:

* Exclusion Criteria Alternate medical or psychiatric illness that explains Long COVID symptoms in the opinion of the Investigator or sub-investigator.

Active or uncontrolled co-morbidities (including depression, untreated endocrine diagnoses), which may interfere with the ability of the patient to participate in the study in the opinion of the Principal Investigator or Sub-Investigator.

Body Mass Index >40 Known allergy to rice flour. Any investigational drug use in the past 30 days. Fatigue improvement because of a current treatment intervention. Treatment within the past 14 days or current treatment with stimulants including methylphenidate, amphetamine-dextroamphetamine, phentermine, lisdexamfetamine, modafinil, and armodafinil Previous or current use of oxaloacetate. Pregnancy, or while breast feeding. Women should not be enrolled within 6 months of giving birth and within 3 months of cessation of breast feeding.

Past medical history of:

Untreated or uncontrolled major depressive disorder, untreated or uncontrolled endocrine diagnoses including hypothyroidism (Hashimoto's, etc.), Grave's disease, adrenal insufficiency, hypogonadism (testosterone deficiency), diabetes mellitus or insipidus.

In the last 3 years have they experienced a concussion with loss of consciousness, brain surgery, an automobile accident with head/neck injury, and/or other traumatic brain injury.

Active supra-ventricular tachycardia or ventricular tachycardia, e.g., atrial fibrillation or flutter, paroxysmal atrial fibrillation, junctional tachycardia, ventricular tachycardia.

Symptomatic hypotension defined as rested sitting systolic BP < 90 mmHg or rested sitting diastolic BP < 60 mmHg, Substance abuse in the past 12 months as determined by self-report or in the opinion of the PI and Sub-I

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Chalder Fatigue Score | 42 days
  A Validated patient derived survey of fatigue

SECONDARY OUTCOMES:
Global Impression of Change | 42 days
  A Validated patient derived survey for overall improvment
Up-Time | 42 days
  Measurement of physical activity with a device attached to the ankle

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda Bateman, MD, Principal Investigator — Bateman Horne Center
Locations (1):
- Bateman Horne Center, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Cash A, Kaufman DL. Oxaloacetate Treatment For Mental And Physical Fatigue In Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) and Long-COVID fatigue patients: a non-randomized controlled clinical trial. J Transl Med. 2022 Jun 28;20(1):295. doi: 10.1186/s12967-022-03488-3. PMID 35764955